CLINICAL TRIAL: NCT03444805
Title: Post-AHSCT (Autologous Hematopoietic Stem Cell Transplantation) Management for Patients With Systemic Sclerosis: a Prospective, Non-interventional Approach Across Europe (NISSC-2) for the Autoimmune Diseases Working Party of the European Group for Blood and Marrow Transplantation (EBMT)
Brief Title: EBMT ADWP Prospective Non-interventional Study: Post-AHSCT Management in SSC Patients (NISSC-2)
Acronym: NISSC-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: ADWP 8410025
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Autoimmune Diseases
Keywords: Autoimmune diseases; Systemic sclerosis; Autologous hematopoietic stem cell transplant (AHSCT); Post-AHSCT management; Immune reconstitution
MeSH Terms: conditions — Autoimmune Diseases; Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NISSC-2: SSC patients treated with AHSCT
  Interventions: Procedure: Autologous HSCT

INTERVENTIONS:
Procedure: Autologous HSCT — 1st AHSCT

SUMMARY:
The aim of the study is to assess the effectiveness of various post-transplant treatment management approaches on clinical and immune biological responses after Autologous Hematopoietic Stem Cell transplantation (AHSCT) for Systemic Sclerosis (SSc) as currently performed by the different treatment protocols used in routine clinical practice across Europe in various EBMT centres

DETAILED DESCRIPTION:
NISSc-2 is a prospective observational study specifically designed to assess the effectiveness of various post-transplant treatment management approaches on clinical and immune biological responses after Autologous Hematopoietic Stem Cell transplantation (AHSCT) for Systemic Sclerosis (SSc) as currently performed by the different treatment protocols used in routine clinical practice across Europe in various EBMT centres through the careful recording and analysis of routinely collected clinical and immune biological data, and specific data regarding post-transplant use of SSc active treatments, including:

* Steroids,
* SSc active treatments after AHSCT such as mycophenolate mofetil (MMF), azathioprine, cyclophosphamide (oral or IV), methotrexate, polyclonal antibodies (such as ATG) or monoclonal antibodies (rituximab, belimumab or any others) as well as their respective dosage and duration of each treatment. These post-transplant treatments can be administered for various reasons, which can be specified by local investigators, such as per local protocol decision for maintenance therapy, or for disease progression with or without prior clinical response, during routine clinical follow-up. Patients who do not receive any post-transplant therapy will also be observed.

Different protocols are used in the different centres, but it is not yet clear, which approach will be the most efficient and the safest. The role of stem cell purification with CD34-selection also needs to be determined prospectively.

In addition, the EBMT Autoimmune Diseases and Immunobiology Working Parties developed and implemented guidelines for 'good laboratory practice' in relation to procurement, processing, storage and analysis of biological specimens for immune reconstitution studies in AD patients before, during and after AHSCT [16]. To follow post-transplant immune reconstitution according to ADWP GCP, results of routine analyses performed by centres under standardized conditions on available biological samples will be investigated in correlation to clinical outcome parameters. Every centre will follow its own local protocol for AHSCT, which usually refers to the recent update of the EBMT guidelines for AHSCT in autoimmune disease.

We therefore specifically designed NISCC-II to prospectively capture various post-ASHCT management protocols and their effect on the observed clinical response after AHSCT.

ELIGIBILITY:
Inclusion Criteria:

1. - Autologous HSCT
2. - Age above 18 years at time of transplant.
3. -. Established diagnosis of progressive SSc according to 2013 ACR/EULAR classification criteria

Exclusion Criteria:

1. Pregnancy or inadequate contraception
2. Severe concomitant disease
3. Reduced lung, cardiac or renal function

   a. .Reduced lung function with FVC < 50% or DLCO < 30% (of predicted values) b; .Pulmonary arterial hypertension with baseline (resting) PASP > 40 mmHg or mPAP > 25 mmHg or a PASP > 45 mmHg or mPAP > 30 mmHg after fluid challenge or Pulmonary vascular resistance > 3 Wood units on RHC c. Severe heart failure with Ejection Fraction < 45% by cardiac echocardiography d. D-sign of septal bounce on cardiac MRI e. Unrevascularized severe coronary artery disease f. Untreated severe arrhythmia g. Cardiac tamponade h. Constrictive pericarditis i. Kidney insufficiency: creatinine clearance <30ml/min Previously damaged bone marrow
   1. Leukopenia < 2.0 x 109/L (total white cell count)
   2. Thrombocytopenia < 100 x 109/L
4. Uncontrolled severe or chronic infection (Hepatitis B/C, HIV, Salmonella carrier, syphilis, tuberculosis)
5. Severe concomitant psychiatric illness (depression, psychosis)
6. Concurrent neoplasms or myelodysplasia in the past 5 years
7. Smoking (current)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated with AHSCT for progressive systemic sclerosis in participating centres
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS), | 2 years post transplant
  defined as survival since AHSCT without evidence of progression of SSc.

SECONDARY OUTCOMES:
Treatment related toxicity | 100 days post-transplant
  Treatment related toxicity throughout the study period using WHO toxicity parameters (expressed as maximum grade toxicity per organ system, see appendix) Incidence of Adverse Events (AE) and Serious Adverse Events (SE) Neutrophil and platelet engraftment, defined as first day after transplantation with absolute neutrophil count > 0.5 x 109/L and platelet count >20 x 109/L (without platelet transfusion).
100 days Treatment Related Mortality (100d TRM) | 100 days post-transplant
  defined as any death during 100 days following transplant that cannot be attributed to progression or relapse of the disease
Overall Survival (OS) | 2 years post-transplant
  Overall survival
Use of prednisone equivalent | 1 year and 2 years post-transplant
  Use of prednisolone equivalent > 6 mg/day for more than 3 months
Use of immunosuppressive drugs | 2 years post-transplant
  defined as use of any post-transplant immunosuppressive drugs (mycophenolate mofetil, azathioprine, oral or iv cyclosphosphamide or methotrexate) for either causes (maintenance therapy as per local protocol decision, SSc progression or relapse) and total duration of exposure to this post-transplant immunosuppressive treatment (average monthly daily dose and months duration)
Use of post-transplant biotherapies | 2 years post-transplant
  defined as use of any monoclonal (i.e. anti CD20, anti-BLyS, alemtuzumab or polyclonal (i.e. ATG) antibodies for either causes (per local protocol decision, EBV infection or reactivation, progression or relapse) and total doses (in number and g/kg)
Response to treatment | 1 year and 2 years post-transplant
  defined as any of the following changes
  * 25% improvement in mRSS and/or
  * ≥10% improvement in DLCO or FVC as compared to baseline (before mobilisation)
Infectious complications, CMV / EBV reactivation | 2 years post-transplant
  Infectious complications, CMV / EBV reactivation
Secondary autoimmune diseases and secondary malignancy | 2 years post-transplant
  defined, autoimmune thrombocytopaenia, autoimmune thyroid disease, autoimmune haemolytic anaemia, Evans' syndrome, acquired haemophila, ulcerative colitis, rheumatoid arthritis and spondyloarthropathy, autoimmune hepatitis, others) and secondary malignancy (EBV lymphoproliferative disorders, AML, MDS, skin cancers, and any others
Immune reconstitution | 2 years post-transplant
  Results of routine analysis performed by centres will be investigated in correlation to clinical outcomes parameters and will allow to follow post-transplant immune reconstitution according to ADWP GCP.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Farge, PhD, Study Chair — EBMT ADWP
Locations (1):
- Badoglio Manuela- EBMT Paris Office, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Organisation website — http://ebmt.org